CLINICAL TRIAL: NCT04370418
Title: Evaluation of the Efficacy and Toxicity of Neo-adjuvant Short Course Radiation Therapy Concurrently With Continuous Infusion 5-fluorouracil in the Management of Locally Advanced Rectal Cancer Patients
Brief Title: Neo-adjuvant Short Course Chemo-radiation Therapy in Locally Advanced Rectal Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mohsen Khalil, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: short course chemoradiation
Record Dates: First submitted 2020-04-25; First posted 2020-05-01 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Neo-adjuvant Short Course Chemo-radiotherapy in Locally Advanced Cancer Rectum
Keywords: CCRTH
MeSH Terms: interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant chemo-radiation (Other): Short-course RT: 5 fractions of 5 Gy to a total dose of 25 Gy over 5 consecutive days. IMRT plans are generated with 6 MV photons.
  Dose-escalated concurrent 5-FU: The 3 doses levels of 5-FU are 100, 150, and 200 mg/m2/d. 5-FU will be given by continuous infusion for 20 hours every day starting on the morning of radiation.
  mFOLFOX: will be given 2 weeks after concurrent chemoradiation for a total of 4 cycles, with each cycle being 14 days. Surgery will be omitted in patients with complete pathological response and proceed to adjuvant chemotherapy. If patient develops progressive or metastatic disease, he/she will be omitted from the investigators study.
  The surgery will be considered 4-8 weeks after end of therapy. Adjuvant mFOLFOX6: 6 cycles chemotherapy will begin between 4 weeks and 8 weeks after surgery.
  Toxicities assessment: be using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
  Interventions: Drug: short course chemo-radiation with 5-fluorouracil

INTERVENTIONS:
Drug: short course chemo-radiation with 5-fluorouracil — neo-adjuvant short course chemo-radiation in locally advanced rectal cancer patients followed by delayed surgery
  Other Names: 5-fu

SUMMARY:
* The primary objective of this trial is to assess the safety and feasibility of 5-FU when given concurrently with5 Gy x 5 fractions IMRT.
* The secondary endpoint is to assess disease local control and the response rate after short course radiotherapy concurrent with dose escalation infusion 5-fu followed by mFOLFOX and delayed surgery.

DETAILED DESCRIPTION:
Neo-adjuvant radiotherapy is associated with the improvement of local control for rectal cancer. For locally advanced stage II-III resectable rectal cancer, either preoperative short-course radiotherapy of 25 Gy in 5 consecutive days or long-course chemo-radiotherapy followed by radical Total Meso-rectal Excision is recommended. The Swedish Rectal Cancer Trial has demonstrated the lower rate of early toxicity of short course radiotherapy when compared to chemo-radiation. Short-course irradiation reduced the risk of local recurrence with evidence of overall survival improvement. Short-course regimen is less expensive and more convenient, especially in centers with long waiting lists. Two meta-analyses showed that short course is as effective as long course chemo-radiation in the management of locally advanced rectal cancer in the terms of sphincter preservation rates, down-staging, R0 resection, local control, and grade 3-4 toxicity. Despite reduction in local-regional recurrence risk with neo-adjuvant short course radiotherapy, distant disease recurrence remains a substantial risk for patients with locally advanced disease. In a controlled randomized trial, a short course radiotherapy followed by consolidation chemotherapy prior to surgery yielded superior overall survival outcomes compared to chemo-radiotherapy, without significant differences in disease-free survival, nor local or distant disease control rates. The phase III RAPIDO and STELLAR clinical trials are also evaluating short course radiotherapy and consolidation chemotherapy. The Stockholm III trial was a 3-arm trial that compared short-course RT with the standard 1-week delay to surgery, short-course RT with a 4- to 6-week delay to surgery, and long-course chemoradiation with a 4- to 6-week delay to surgery. The results show similar outcomes between the groups, but delaying the surgery after short-course RT decreased the rates of high-grade toxicity and allowed for an expedited treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed cancer rectum
* Age between 20-80
* Clinical T3\4 or node positive disease by MRI

Exclusion Criteria:

* Early stage cancer rectum
* M1 disease confirmed by imaging or pathological

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment adverse events as assessed by National Cancer Institute Common Terminology Criteria for adverse events version 4.0 | baseline
  Dose limiting toxicity is defined as any of the following occurring during chemo radiation or within 21 days from the completion of the treatment like grade 4 non hematological toxicity, grade 4 febrile neutropenia, grade 4 thrombocytopenia or neutropenia toxicity lasting 7 days, grade 3 non hematological toxicity preventing treatment more than 3 days, elevation of ALT or AST more than 10 the upper limit of normal for 7 days

SECONDARY OUTCOMES:
assess disease local control and the response rate after short course radiotherapy concurrent with dose escalation infusion 5-fu followed by mFOLFOX and delayed surgery. | 2 years
  assess disease local control measured by disease free survival in months and the response rate after short course radiotherapy concurrent with dose escalation infusion 5-fu followed by mFOLFOX and delayed surgery measured by either complete pathological response 0r partial response or no response

CONTACTS AND LOCATIONS:
Overall Officials: taha z mohran, professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trakarnsanga A, Ithimakin S, Weiser MR. Treatment of locally advanced rectal cancer: controversies and questions. World J Gastroenterol. 2012 Oct 21;18(39):5521-32. doi: 10.3748/wjg.v18.i39.5521. PMID 23112544
- [Background] Swedish Rectal Cancer Trial; Cedermark B, Dahlberg M, Glimelius B, Pahlman L, Rutqvist LE, Wilking N. Improved survival with preoperative radiotherapy in resectable rectal cancer. N Engl J Med. 1997 Apr 3;336(14):980-7. doi: 10.1056/NEJM199704033361402. PMID 9091798
- [Background] Bujko K, Nowacki MP, Nasierowska-Guttmejer A, Michalski W, Bebenek M, Kryj M. Long-term results of a randomized trial comparing preoperative short-course radiotherapy with preoperative conventionally fractionated chemoradiation for rectal cancer. Br J Surg. 2006 Oct;93(10):1215-23. doi: 10.1002/bjs.5506. PMID 16983741
- [Background] Zhou ZR, Liu SX, Zhang TS, Chen LX, Xia J, Hu ZD, Li B. Short-course preoperative radiotherapy with immediate surgery versus long-course chemoradiation with delayed surgery in the treatment of rectal cancer: a systematic review and meta-analysis. Surg Oncol. 2014 Dec;23(4):211-21. doi: 10.1016/j.suronc.2014.10.003. Epub 2014 Oct 29. PMID 25466851
- [Background] Kairevice L, Latkauskas T, Tamelis A, Petrauskas A, Pauzas H, Zvirblis T, Jarusevicius L, Saladzinskas Z, Pavalkis D, Janciauskiene R. Preoperative long-course chemoradiotherapy plus adjuvant chemotherapy versus short-course radiotherapy without adjuvant chemotherapy both with delayed surgery for stage II-III resectable rectal cancer: 5-Year survival data of a randomized controlled trial. Medicina (Kaunas). 2017;53(3):150-158. doi: 10.1016/j.medici.2017.05.006. Epub 2017 Jun 22. PMID 28690144
- [Background] Bujko K, Wyrwicz L, Rutkowski A, Malinowska M, Pietrzak L, Krynski J, Michalski W, Oledzki J, Kusnierz J, Zajac L, Bednarczyk M, Szczepkowski M, Tarnowski W, Kosakowska E, Zwolinski J, Winiarek M, Wisniowska K, Partycki M, Beczkowska K, Polkowski W, Stylinski R, Wierzbicki R, Bury P, Jankiewicz M, Paprota K, Lewicka M, Cisel B, Skorzewska M, Mielko J, Bebenek M, Maciejczyk A, Kapturkiewicz B, Dybko A, Hajac L, Wojnar A, Lesniak T, Zygulska J, Jantner D, Chudyba E, Zegarski W, Las-Jankowska M, Jankowski M, Kolodziejski L, Radkowski A, Zelazowska-Omiotek U, Czeremszynska B, Kepka L, Kolb-Sielecki J, Toczko Z, Fedorowicz Z, Dziki A, Danek A, Nawrocki G, Sopylo R, Markiewicz W, Kedzierawski P, Wydmanski J; Polish Colorectal Study Group. Long-course oxaliplatin-based preoperative chemoradiation versus 5 x 5 Gy and consolidation chemotherapy for cT4 or fixed cT3 rectal cancer: results of a randomized phase III study. Ann Oncol. 2016 May;27(5):834-42. doi: 10.1093/annonc/mdw062. Epub 2016 Feb 15. PMID 26884592
- [Background] Nilsson PJ, van Etten B, Hospers GA, Pahlman L, van de Velde CJ, Beets-Tan RG, Blomqvist L, Beukema JC, Kapiteijn E, Marijnen CA, Nagtegaal ID, Wiggers T, Glimelius B. Short-course radiotherapy followed by neo-adjuvant chemotherapy in locally advanced rectal cancer--the RAPIDO trial. BMC Cancer. 2013 Jun 7;13:279. doi: 10.1186/1471-2407-13-279. PMID 23742033
- [Background] J. Jin YT, S. Liu, Y. Zhu, W. Wang, G. Li, X. Wang, J. Wang, J. Yang, S. Li, N. Li, W. Liu, Y. Li, Y. Chi, A. Zhou, J. Huang, X. Wang, L. Jiang, J. Jiang, S. Zou. Short-term radiotherapy plus chemotherapy versus long-term chemoradiotherapy in locally advanced rectal cancer (STELLAR): a planned interim analysis. Annals of Oncology. 2018;29(suppl 8):167.
- [Background] Erlandsson J, Holm T, Pettersson D, Berglund A, Cedermark B, Radu C, Johansson H, Machado M, Hjern F, Hallbook O, Syk I, Glimelius B, Martling A. Optimal fractionation of preoperative radiotherapy and timing to surgery for rectal cancer (Stockholm III): a multicentre, randomised, non-blinded, phase 3, non-inferiority trial. Lancet Oncol. 2017 Mar;18(3):336-346. doi: 10.1016/S1470-2045(17)30086-4. Epub 2017 Feb 10. PMID 28190762
- [Background] Wu H, Fang C, Huang L, Fan C, Wang C, Yang L, Li Y, Zhou Z. Short-course radiotherapy with immediate or delayed surgery in rectal cancer: A meta-analysis. Int J Surg. 2018 Aug;56:195-202. doi: 10.1016/j.ijsu.2018.05.031. Epub 2018 May 25. PMID 29807169